CLINICAL TRIAL: NCT01801514
Title: Applications of Dual-Energy Computed Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: iCT DL
Record Dates: First submitted 2013-02-27; First posted 2013-02-28 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Other Conditions That May Be A Focus of Clinical Attention
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Computed Tomography scan — Routine Computed Tomography scan

SUMMARY:
The purpose of the study is to evaluate the feasibility of multilayer detection-based dual energy computed tomography scanner and to assess the added diagnostic value of dual energy applications

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject
2. Subjects with relative clinical findings indicative for CT examination. CT referral request approved by a physician is needed
3. Voluntary signed the Informed Consent Form

Exclusion Criteria:

1. Pregnant or potentially pregnant female subjects
2. Subjects who are not able or not willing to give written Informed Consent without a caregiver consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Capability of producing dual energy computed tomography imaging and dual energy applications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sosna, MD, Principal Investigator
Locations (1):
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel